CLINICAL TRIAL: NCT06555900
Title: Predicting Episodes of Intracranial Hypertension in Neuro-injured Patients: Development of a Decision Algorithm Using Artificial Intelligence
Brief Title: Predicting Episodes of Intracranial Hypertension in Neuro-injured Patients: Development of a Decision Algorithm Using Artificial Intelligence (PREDICT-CE)
Acronym: PREDICT-CE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0293 - PREDICT-CE
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Creation of a Warehouse of Clinical Data and Physiological Signals at the Patient's Bedside

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators wish to build up a database of clinical data and physiological signals with a view to developing a predictive algorithm based on continuous analysis of the intracranial pressure waveform and other parameters commonly used in intensive care to predict the occurrence of an episode of intracranial hypertension (HTIC). This algorithm will be designed using supervised learning statistical methods based on innovative statistical analysis methods (artificial intelligence). These methods are classically used to exploit massive data such as sensor data.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years
* admission to intensive care for less than 3 days for a neurological lesion
* Sensor placement for intracranial pressure monitoring

Exclusion Criteria:

* patient under judicial protection
* refusal to participate
* patients under 18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any neuro-injured patient admitted to intensive care
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Creation of a database of clinical data and physiological signals to develop a predictive algorithm based on continuous analysis of the intracranial pressure waveform to predict the occurrence of an episode of intracranial hypertension. | 30 minutes
  Occurrence of an episode of intracranial hypertension defined as ICP >20mmHg for 30 minutes

SECONDARY OUTCOMES:
Predict long-term functional outcome using intracranial pressure wave signal modeling and other parameters collected in real time | 28 days
  Occurrence of vasospasm diagnosed by cerebral perfusion angioscanner

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three month and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.